CLINICAL TRIAL: NCT07223931
Title: Clinical Validation of the Dozee System for Contactless Monitoring of Heart Rate, Respiration Rate, Motion, and Bed-Exits
Brief Title: Validating Dozee for Contactless Monitoring of Heart, Breathing, and Movemen
Status: Recruiting | Type: Observational
Sponsor: Turtle Shell Technologies Pvt. Ltd. (Industry)
Collaborators: Eastside Research Associates (Unknown)
Responsible Party: Sponsor
Other Study IDs: DZ_VS_VAL
Record Dates: First submitted 2025-09-23; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: No Specific Medical Conditions or Disease States; No Specific Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Arm Study (Cohort): Group/Cohort Description: All participants will be on standard telemetry monitoring for Heart Rate and Respiration Rate using the gold standard (Electrocardiography and Capnography respectively). In addition, a contactless monitoring devices will be placed on the patient bed to measure data. This device is Dozee VS (Investigational Device). Data from all devices will be measured simultaneously.
  Interventions: Device: Device: Telemetry monitoring

INTERVENTIONS:
Device: Device: Telemetry monitoring — All participants will be on standard telemetry monitoring for Heart Rate, Respiration Rate and movements using the gold standard (Electrocardiography and Capnography respectively).

SUMMARY:
The Dozee VS system (K221555) is a contactless device that tracks heart rate and breathing rate using a sensor sheet placed under the mattress. It captures body vibrations and converts them into vital signs, which can be monitored remotely in real time. The system also supports add-ons like a blood pressure cuff, pulse oximeter, and thermometer, offering a complete monitoring solution. This study aims to validate the updated AI-powered heart rate and improved breathing rate algorithms across different sensor sheet types to confirm clinical accuracy

DETAILED DESCRIPTION:
The Dozee VS system (K221555), developed by Turtle Shell Technologies, is a non-invasive, contactless device that continuously monitors heart rate (HR) and breathing rate (RR). A thin sensor sheet placed under the mattress detects tiny body vibrations from the heart and lungs, which are processed by smart algorithms and displayed on a secure online dashboard for real-time monitoring.

Unlike traditional methods such as ECGs, nasal tubes, or thermistors-which are invasive, require skilled placement, and are uncomfortable for long-term use-Dozee is simple, comfortable, and doesn't rely on patient compliance like wearables do. The system can also connect to add-on devices, including a blood pressure cuff, pulse oximeter, and thermometer, giving a full picture of a patient's vital signs and helping spot early signs of deterioration.

Hardware upgrades now include dual-sensor sheets that improve accuracy across different mattresses and patient types. The new HR algorithm uses AI/ML for better accuracy, while the improved RR algorithm performs more reliably even with movement or weak signals.

Study Goal: This study aims to validate the updated algorithms (Gen 2) for HR and RR across the three sensor sheet types (DS, S1, and S1-I) to ensure they meet clinical accuracy standards

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if they meet the following inclusion criteria:

1. Adults Male or female. (Above 18 years of age)
2. Provide written informed consent.
3. Weight between 40kg/88.18lbs and 120kg/264.55lbs
4. Agree to not eat during the testing period
5. Able to move and exit the bed independently and safely.

Exclusion Criteria:

Subjects will be excluded if they have any of the following inclusion criteria:

1. Are connected to a device that may interfere with the device monitoring in this study.
2. Are receiving any bedside care which may be incompatible with the study procedures.
3. A likely need to receive or undergo a procedure during the testing period.
4. Cannot accept a nasal cannula, or have an ECG leads placed on the chest.
5. Have a significant medical condition in the judgement of the investigator, which may compromise the study testing procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on atleast 60 subjects in the age group above 18 years regardless of gender. The patients/volunteers be informed about the study and a written informed consent form will be obtained from them. Dozee will be placed under the mattress of the patient's bed and the data will be collected through the device whenever a patient is on the bed.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Absolute Error (MAE) of Dozee's Heart Rate a from the Gold Standard ECG | 6 months
  Heart Rate collected at 1 Min intervals from gold standard and Dozee. Mean Absolute Error (MAE) of the Dozee Heart Rate will be calculated.
Accuracy (%) of Dozee in identfying subject movement | 6 months
  Time stamps of subject movement during the study will be recorded manullay. Time stamps of Dozee's movement will be recorded. Accuracy of the Dozee device in detecting movement compared to manual observation will be computed in terms of percentage.
Accuracy(%) of of Dozee's bed-exits | 6 months
  Time stamps of bed-exits will be recorded manually during the study will be recorded. Time stamps of Dozee's bed-exit will be computed. Accuracy of the Dozee device in detecting bed-exit compared to manual observation as gold standard will be computed in terms of percentage.
Mean Absolute Error (MAE) of Dozee's Respiratory Rate from the Gold Standard Capnography | 6 Months
  Respiratory Rate collected at 1 Min intervals from gold standard and Dozee. Mean Absolute Error (MAE) of the Dozee Respiratory Rate will be calculated.

SECONDARY OUTCOMES:
Range of values (minimum, maximum, and spread) of Heart Rate in beats per min measured by the gold standard and the Dozee | 6 months
  The outcome will be assessed by comparing the range of values (minimum, maximum, and spread) of Heart Rate ( beats per minute) measured by the gold standard and the Dozee over the study period.
Range of values (minimum, maximum, and spread) of Respiratory Rate in breaths per min measured by the gold standard and the Dozee | 6 Months
  The outcome will be assessed by comparing the range of values (minimum, maximum, and spread) of Respiratory Rate ( breaths per minute) measured by the gold standard and the Dozee over the study period.
Bland- Altman Level of Agreement between Dozee Heart Rate and Respiratory Rate with the Gold Standard | 6 months
  Level of Agreement between Dozee's HR and RR with reference device computed by Bland Altman.
Detection rate (%) of the Dozee's Heart Rate and Respiratory Rate | 6 months
  The time-stamps of Dozee's Heart Rate and Respiratory Rate and the gold standard Heart Rate and Respiratory Rate will be recorded. DR is the proportion of gold standard points for which the DS successfully provides a corresponding measured value, relative to the total number of gold standard points.
Level of Agreement between Dozee Heart Rate and Respiratory Rate with the Gold Standard | 6 months
  Level of Agreement between Dozee Heart Rate and Respiratory Rate with the Gold Standard by using Deming Regression with Pearson Co-efficient

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Chilka, MD, Principal Investigator — ERA Health Research
Locations (1):
- ERA Health Research, Midland, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) are protected under HIPPA Act of 1996.